CLINICAL TRIAL: NCT02812615
Title: Stunting and Bangladesh Environmental Enteric Dysfunction Study
Brief Title: The Bangladesh Environmental Enteric Dysfunction Study
Acronym: BEED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); University of Virginia (Other); University of Washington (Other); Dhaka Medical College (Other); Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PR-16007
Record Dates: First submitted 2016-05-31; First posted 2016-06-24 (Estimated); Last update posted 2022-02-11 (Actual); Status verified 2021-12

CONDITIONS: Malnutrition; Infection
Keywords: Environmental Enteric Dysfunction
MeSH Terms: conditions — Malnutrition; Infections | interventions — Eggs; Milk; Albendazole; Pyrantel Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Malnourished participants (Experimental): After screening the participants for any organic diseases and application of inclusion/exclusion criteria, stunted children, children who are at risk of stunting and malnourished adult cases will receive one egg, 150 ml of milk 6 days a week for 3, 2 and 2 months respectively. Along with that participants will also get Anti-helminthic treatment (Albendazole/Pyrantel Pamoate) and nutritional counselling. Children will get one sachet of multiple micro-nutrient sprinkles per day to be administered at home with the mid-day meal for two months.
  Interventions: Dietary Supplement: Egg; Dietary Supplement: Milk; Drug: Albendazole/Pyrantel Pamoate; Behavioral: Nutritional counselling; Dietary Supplement: Micronutrient sprinkles

INTERVENTIONS:
Dietary Supplement: Egg — After enrollment, participants will receive one large egg 6 days a week for 3, 2 and 2 months for stunted children, children at risk of stunting, and malnourished adults, respectively.
Dietary Supplement: Milk — After enrollment, participants will receive 150ml of milk 6 days a week for 3, 2 and 2 months for stunted children, children at risk of stunting, and malnourished adults, respectively.
Drug: Albendazole/Pyrantel Pamoate — As per the national guidelines, treatment will be provided based with 200 mg of Albendazole or 10mg/kg Pyrantel Pamoate single dose if the participants have not been treated for helminths in the preceding three months.
Behavioral: Nutritional counselling — Parents/caregivers will be given nutritional counselling
Dietary Supplement: Micronutrient sprinkles — For the child cohort, one sachet of multiple micro-nutrient sprinkles per day to be administered with the mid-day meal for two months

SUMMARY:
This is a community-based intervention study which will be undertaken at Mirpur, Dhaka, Bangladesh. Participants will be recruited from two age groups: a child cohort (age 12 to 18 months) and an adult cohort (age 18 to 45 years). The child cohort will consist of stunted children (length for age Z score, LAZ < -2), children who are at risk of stunting (length for age Z score <-1 to -2) and child controls. The adult cohort will consist of malnourished adult cases (Body Mass Index <18.5) and adult controls. After screening the participants for any organic diseases and application of inclusion/exclusion criteria, they will receive nutrition interventions. Participants eligible for study will be tested for potential bio markers of environmental enteropathy (stool, urine and serum) once before and once after the nutritional intervention. Participants who will fail to respond to nutritional therapy (measured by anthropometric assessment) will become candidates for upper gastrointestinal endoscopy with biopsy. The study will include duodenal biopsies from a control group of children from University of Virginia Hospital in Charlottesville, Virginia who will undergo upper GI endoscopy as part of their clinical care as per the standard clinical protocol followed at the hospital. Adult controls (BMI > 18.5) for endoscopy will be collected from international centre for diarrhoeal disease research,Bangladesh staff clinic, Dhaka Medical College and Hospital (DMCH), Dhaka and Bangabandhu Sheikh Mujib Medical University (BSMMU), Dhaka.

DETAILED DESCRIPTION:
Study design This will be a community-based intervention study. Survey, screening, enrollment of subjects will be done in Mirpur in Dhaka city.

Subjects Participants will be recruited from two age groups: a child cohort (age 12 to 18 months) and an adult cohort (age 18 to 45 years). The child cohort will consist of two groups of children- stunted children (LAZ score < -2) and children who are at risk of stunting (LAZ <-1 to -2). A group of malnourished adults (BMI <18.5) will also be enrolled from the parents of children and by a cross sectional survey from Mirpur area of Dhaka city.

Sample size:

Participants will be collected and recruited in a cross sectional manner. Based on a sample size calculation with 10% precision and 95% confidence interval, a minimum of 35 stunted children, 35 at risk of stunting children and 35 adults will be recruited. So, the final sample size for endoscopy is 105 subjects (35+35+35). As endoscopy is an invasive procedure, it was assumed that only one-third of those who would fail to respond after nutrition intervention would give consent for endoscopy. So, basic sample size was increased three times for a minimum of 105 (35 x 3) stunted children (LAZ <-2), 105 (35 x 3) children at risk of stunting (LAZ <-1 to 2) and 105 (35 X 3) malnourished adults (BMI < 18.5) who would fail to thrive. To achieve that 525 stunted children, 525 children at risk of stunting and 525 malnourished adults for nutrition interventions will be recruited as it was assumed that ~20% of each group will fail to respond despite the nutritional intervention. For that order of recruitment surveying at least 3977 (1312+2665) children 12-18 months old and 2100 adults based on the current prevalence of malnutrition in the two age groups is required. For adult control group, same number (35) of adult controls will be recruited from Dhaka Medical College and international centre for diarrhoeal disease research,Bangladesh staff clinic by convenient sampling method

Description of field site:

The study will be conducted among residents of Mirpur, one of the 21 administrative units of the nation's capital, Dhaka.

Recruitment, Screening and Consenting If the participants are interested to volunteer in the study, the designated staff will proceed to screening and consenting. Screening will consist of a review of the inclusion and exclusion criteria listed above. If the subject is eligible to participate, the process will proceed to consenting consisting of a thorough review of the written consent form in a manner appropriate for the child's parents' / participants literacy level. Prior to signing the consent form, they will have an opportunity to ask any questions about the study. If the Field Research Assistant (FRA) determines that participants have demonstrated adequate comprehension of the study, the consent form will be signed by the FRA and the child's parent(s) /adult participants. If the parent(s) / adult participants are not sufficiently literate to read and/or sign the consent form, consenting and a thumb impression will be obtained in the presence of a witness who is not associated with the study. The child's parent(s) / adult participants will be provided with a copy of the signed consent form.

Detailed procedure of Directly Observed Nutritional Therapy:

After enrollment, participants will receive daily directly observed nutritional therapy. Nutritional therapy consists egg and milk and will be provided by the study free of cost. Duration of nutrition interventions will be 3, 2 and 2 months for stunted children, children at risk of stunting, and malnourished adults, respectively and nutritional therapy will be delivered between the morning and mid day meal, anytime between 10:00 am to 11:30 am. Participants will be asked to come to the designated nutrition center (to be established at Mirpur) daily for nutritional therapy to avoid the issue of food sharing. A staff will visit the family's household if a participant defaults in coming to the nutrition center. In addition to the food based nutritional therapy, participants will receive the following nutritional and health support:

* Anti-helminthic treatment (Albendazole/Pyrantel Pamoate) as per national guidelines
* Parents/caregivers will be given nutritional counselling
* For the child cohort, parents will be given one sachet of multiple micro-nutrient sprinkles per day for two months.
* Any inter-current illnesses detected by the study team will also be taken care of.

Food based nutritional therapy: Supplementation of the usual home diet with one egg, and 150 ml of whole milk which will provide an additional 178 kilo-calories, 11.1 g protein, and 11.5 g of fat to the daily diet of enrolled subjects. Sachets of multiple micro-nutrient powder will be provided for use at home at dinner.

In order to clarify the role of food-based nutritional therapy, there will be comparison subgroups of 40 stunted children and 40 children at risk of stunting who will be followed for 3 and 2 months respectively, without any nutritional therapy. At the end of the observation period of 3 and 2 months, nutritional therapy will be provided to these children same as that provided to the enrolled participants.

Discontinuation from the study: A child will be discontinued from the study and referred for medical evaluation if he/she shows reluctant to feed for consecutive 7 days which includes daily intake of 50% or less amount of food that will be offered. A new eligible child will be recruited in his position for nutritional intervention.

Collection of biological samples:

All biological samples (blood, urine, stool, duodenal aspirates, and endoscopic biopsies) will be collected as per the standard operative procedures (SOPs) which will be prepared for this protocol. A total amount of 5ml blood will be collected from each participant before and after nutritional intervention. Urine will be collected for Lactulose-Rhamnose assay, and for metabolomic studies; breath samples will be collected for testing for small intestinal bacterial overgrowth (SIBO). Second SIBO will be done 1-2 weeks prior to endoscopy so that the findings from the endoscopy can be compared to the breath tests. Fecal samples will be collected for biomarkers, Taqman array card (TAC) assays and Microbiome/Microbiota for age Z-score (MAZ)/Bug fluorescence-activated cell sorting.

Detailed procedure of Bio-marker testing

The bio-markers going to be tested for are-

Stool bio-markers

* Regeneration gene 1Beta
* Neopterin
* Myeloperoxidase
* Alpha-1-antitrypsin
* Calprotectin
* The TaqMan Array Card for enteropathogen
* Gut Microbiome analysis
* Bug Fluorescence-Activated Cell Sorting.

Urine bio-markers

• Lactulose-Rhamnose test

Blood bio-markers

* C- Reactive Protein
* Alpha-1-acid glycoprotein
* Soluble cluster of differentiation 14
* Kynurenine-Tryptophan Ratio
* Glucagon-like peptide-2
* Insulin-like growth factor-2
* Tissue Transglutaminase
* Ferritin
* Zinc
* Pepsinogen I/II Ratio
* Low density lipoprotein related receptor 1 (LRP1)
* Blood plasma metabolomics

Other proposed biomarkers

• Small intestinal bacterial overgrowth

After completion of nutritional therapy, all enrolled participants will have an assessment for response which will include:

* Anthropometric measurements
* Collection of one 5 ml blood sample for serum bio-markers of gut function and screening tests for the endoscopy with biopsy procedure, if the procedure is indicated for failure to thrive
* Collection of stool specimen for bio-markers of gut function
* Administration of lactulose-rhamnose solution and collection of urine for up to 2 hours for urine bio markers of gut function

At this time, the final inclusion criterion for endoscopy with biopsy will be evaluated to determine whether the participants failed nutritional therapy or had an adequate response, or have an underlying disease that caused the malnutrition. Failure of nutritional therapy in this study, or failure to respond, is defined in the absence of any other underlying diseases such as tuberculosis:

* LAZ score remains < -2 for stunted children cohort
* LAZ score remains < -1 for "at risk of stunting" children cohort
* BMI < 18.5 and < 10% increase in BMI for adults.

Participants who meet the study definition of "failure to respond" will be checked for presence of any secondary cause of malnutrition like tuberculosis, carcinoma, any parasitic infection etc. Stool microscopy for parasite identification will be done at icddr,b parasitology lab as soon as possible after collection of stool samples. If nothing conclusive can be found, the participants may be requested to undergo preparations for upper GI endoscopy with biopsy, as they may benefit from further evaluation to identify the potential cause(s) of intervention failure and to determine an appropriate therapeutic course. It will also benefit others by validating the non-invasive bio-marker signature of Environmental Enteric Dysfunction. Participants who will undergo endoscopy will receive necessary treatments according to diagnosis.

Participants having celiac disease and clotting disorder (tested by prothrombin time / International Normalized Ratio coagulopathy) will be excluded from the study. Endoscopy of upper gastrointestinal tract will be done as per standards recommended by North American Society for Pediatric Gastroenterology, Hepatology and Nutrition (NASPGHAN0, American College of Gastroenterology (ACG) and American Society for Gastrointestinal Endoscopy (ASGE).

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for stunted children: All of the following criteria must be met for a subject to be eligible to participate in the study-

* Parent(s) willing to sign consent form
* Child age 12-18 months
* LAZ < -2
* Parent(s) willing to bring child to the study site every day for 3 months for nutritional therapy
* Parents willing to have child undergo laboratory investigations and upper GI endoscopy and biopsy if the child fails to respond to nutritional therapy

Inclusion criteria for children who are at risk of stunting: All of the following criteria must be met for a subject to be eligible to participate in the study -

* Parent(s) willing to sign consent form
* Child age 12-18 months
* LAZ between <-1 to -2
* Parent(s) willing to bring child to the study site every day for 2 months for nutritional therapy
* Parents willing to have child undergo endoscopy and biopsy if the child fails to respond to nutritional therapy

Inclusion criteria for malnourished adults: All of the following criteria must be met for a subject to be eligible to participate in the study -

* Willing to sign consent form
* Age 18-45 years
* BMI < 18.5
* Willing to visit the study site every day for 2 months for nutritional therapy
* Willing to undergo endoscopy and biopsy if he/she fails to respond to nutritional therapy

Selection criteria for adult controls:

An equal number of age and sex matched adult controls will be enrolled form the subjects with functional dyspepsia (FD) with apparently normal health (normal BMI) and absence of organic diseases. FD subjects will be identified from the Gastroenterology outpatient department of Dhaka Medical College Hospital and international centre for diarrhoeal disease research, Bangladesh staff clinic who will undergo upper GI endoscopy for evaluation of dyspepsia and have normal endoscopic findings. Dyspepsia will be defined by pre-defined criteria (Rome III criteria) by a structured questionnaire which has been translated and validated in Bengali.

Exclusion Criteria:

Exclusion criteria for stunted children: Meeting any of the following criteria will exclude a subject from study participation -

* Severe acute malnutrition (SAM), severe anemia (<8 g/dl), tuberculosis, other chronic diseases or any congenital disorder or deformity
* Diarrhoea: Ongoing episode of diarrhoea, history of persistent diarrhoea in the past month or history of acute diarrhoea in the past 7 days
* Known allergy to eggs or milk or milk intolerance

Exclusion criteria for children who are at risk of stunting: Meeting any of the following criteria will exclude a subject from study participation -

* Severe acute malnutrition (SAM), severe anemia (<8 g/dl), tuberculosis, other chronic diseases or any congenital disorder or deformity
* Diarrhoea: Ongoing episode of diarrhoea, history of persistent diarrhoea in the past month or history of acute diarrhoea in the past 7 days
* Known allergy to eggs or milk or milk intolerance

Exclusion criteria for malnourished adults: Meeting any of the following criterions will exclude a subject from study participation-

* Severe anemia (<8 g/dl), tuberculosis and other chronic diseases including diabetes mellitus or any congenital disorder or deformity
* Pregnant women, lactating women, drug abusers, known psychiatric disorders
* High clinical suspicion of cancer or other chronic or acute diseases that may cause malnutrition. Adult participants who fulfilled the inclusion criteria and not excluded through history and clinical examination based exclusion criteria will undergo screening tests for confirmation.

Ages: 12 Months to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1575 (Estimated)
Dates: Start 2016-07-16 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Length for Age Z score | baseline and 3 months
  For stunted child participants, length and age data will be collected before and after the intervention period (3 months) and changes in length for age Z score will be measured.For at risk of stunting child participants, length and age data will be collected before and after the intervention period (2 months) and changes in length for age Z score will be measured.
Change in Body Mass Index | baseline and 2 months
  For malnourished adult participants, height and and weight data will be collected before and after the intervention period (2 months) and changes in Body Mass Index will be measured.

SECONDARY OUTCOMES:
Change in stool Regeneration gene 1 Beta (Reg 1B) biomarker level | baseline and 3 months
  Reg1 is known to promote intestinal epithelial cell proliferation, regeneration and repair, and is up-regulated in a variety of enteric infections and inflammatory conditions. A commercial ELISA assay will be run on fecal samples to measure Reg 1 levels.
Change in stool neopterin level | baseline and 3 months
  Neopterin is a product of the breakdown of cyclic guanosine monophosphate (cGMP) when released from phagocytic cells, and an increase in neopterin can be found with the activation of cellular immune response. So, increased neopterin in stools will be used as a marker for an inflammatory immune response in the intestinal epithelium.
Change in stool myeloperoxidase level | baseline and 3 months
  Derived from azurophil granules, which are a specific marker of polymorphonuclear leukocytes (PMN) activity, myeloperoxidase (MPO) catalyzes the oxidation of substances through hydrogen peroxide (H2O2). The MPO H2O2-system has a toxic effect on many micro-organisms such as bacteria, fungi, viruses and mycoplasma. MPO determination in the stool reflects the inflammatory activity of Crohn's disease or ulcerative colitis. During inflammation in the intestinal mucosa, neutrophils migrate towards the gut mucosa and release myeloperoxidase from granulocytes which can be detected in stools and used as a marker of intestinal inflammation. A commercial ELISA kit will be used to measure myeloperoxidase in stool specimens.
Change in stool Alpha-1-antitrypsin level | baseline and 3 months
  Alpha-1-antitrypsin is an acute phase protein predominantly made in the liver, but also in intestinal macrophages, monocytes, and epithelial cells and released during inflammation. The presence of alpha-1-antitrypsin in the stool is a marker of intestinal inflammation, intestinal permeability and protein loss. A commercial ELISA kit will be utilized to measure alpha-1-antitrypsin in stool specimens.
Change in stool Calprotectin level | baseline and 3 months
  Calprotectin is released by activated neutrophils, and it accounts for more than 40% of the cytosolic proteins of neutrophils. Elevated concentrations of calprotectin can be measured in plasma, cerebrospinal fluid, synovial fluid, urine, and feces when inflammation is present or in malignant conditions. The high fecal calprotectin concentrations can be explained by increased turnover of leukocytes in the gut wall and increased migration of neutrophils into the gut lumen . The fecal calprotectin results are expressed in mg of calprotectin per kilogram of wet feces within a normal reference range of <50 mg/kg.
Change in stool TaqMan Array Card (TAC) result | baseline and 3 months
  The TaqMan Array Card (TAC) system is a real-time polymerase chain reaction format that is used to detect multiple infection targets. An enteric TaqMan Array Card can detect 27 enteropathogens, including viruses and helminths Fecal samples will be spiked with extrinsic controls, and total nucleic acid will be extracted. TAC allows fast, accurate, and quantitative detection of a broad spectrum of enteropathogens.
Change in gut microbiota maturity status | baseline and 3 months
  The human gut microbiota undergoes a defined postnatal developmental program of assembly over the first 2-3 years of life that is perturbed in children with undernutrition and is not durably repaired by existing therapeutic foods. While these studies have identified a link between microbiota maturity and anthropometric measures of healthy growth in early childhood, the relationship between histopathologically defined Environmental Enteric Dysfunction and the configuration/maturation of the microbiota in the small and large intestines has not been studied.
Change in lactulose and rhamnose permeability test | baseline and 3 months
  The lactulose and rhamnose permeability test will be used to measure intestinal permeability. The synthetic disaccharide, lactulose, is minimally absorbed via the paracellular route and then excreted unchanged in the urine, while the monosaccharide sugar rhamnose, being smaller is usually completely absorbed in the small intestine and excreted unchanged in the urine. An elevated lactulose: rhamnose ratio indicates increased permeability.
Change in blood C-reactive protein level | baseline and 3 months
  C-reactive protein (CRP) is an acute phase protein and can be detected during infection. It is a measurement of enteric permeability across the gut membrane. A commercial ELISA kit will be used to measure the levels of CRP in plasma samples.
Change in blood Alpha-1-acid glycoprotein level | baseline and 3 months
  Alpha-1-acid glycoprotein is an acute phase protein. Increased levels are found in the serum during systemic tissue injury, inflammation and infection. A commercial ELISA kit will be utilized to measure the levels of alpha-1-acid glycoprotein in plasma specimens.
Change in blood sCD14 level | baseline and 3 months
  sCD14 is a protein receptor for lipopolysaccharide (LPS). Similar to the principle behind the anti-LPS antibody assay, once the LPS or endotoxin containing particles enters the bloodstream from the intestinal mucosa, they are bound to sCD14. An increase in sCD14 indicates an increase in endotoxin or LPS entering the bloodstream from the intestinal mucosa .
Change in blood kynurenine Tryptophan ratio | baseline and 3 months
  Tryptophan is an essential amino acid that is central to cellular respiration and neurotransmission, and is a key immune mediator. During inflammation, tryptophan is metabolized by indoleamine 2,3-dioxygenase (IDO) to the toxic metabolite kynurenine. IDO activity is measured by the ratio of kynurenine to tryptophan. IDO activity correlates with disease severity in patients with chronic inflammatory diseases .
Change in blood Glucagon-like peptide-2 level | baseline and 3 months
  Glucagon-like peptide-2 (GLP-2) is a newly discovered gastrointestinal peptide with 33% sequence homology to glucagon. GLP-2 has attracted interest because of its potent endocrine/paracrine actions. The peptide results from expression of the glucagon gene in the intestinal mucosa, from where it is released mainly in response to luminal contact with unabsorbed nutrients. In addition to mucosal growth, GLP-2 enhances activities of several intestinal brush-border enzymes, and it delays gastric transit, thereby increasing the intestinal capacity for nutrient absorption. Thus, it appears that GLP-2 serves to ensure an optimal intestinal capacity.
Change in blood ferritin level | baseline and 3 months
  Serum ferritin is widely recognized as an acute phase reactant and marker of acute and chronic inflammation, and is nonspecifically elevated in a wide range of inflammatory conditions.
Change in blood zinc level | baseline and 3 months
  Scientists have explored the overlapping nature of zinc deficiency and environmental enteropathy, and presented evidence for their interaction. Environmental Enteropathy (EE) leads to impaired zinc homeostasis, predominantly due to reduced absorptive capacity arising from disturbed intestinal architecture, and zinc deficiency exacerbates several of the proposed pathways that underlie EE, including intestinal permeability, enteric infection, and chronic inflammation.
Change in blood pepsinogen I & II level | baseline and 3 months
  Gastric acid has an important pathophysiological role in human beings. Appropriate levels of gastric acid are needed to adequately absorb many nutrients including minerals and vitamins. It is also a crucial part of the immune system. The hypochlorhydria induced by H. pylori infection may also result in alterations in the gut microbiota and contribute to small intestinal permeability changes and malabsorption,In this study, we also want to investigate serum pepsinogen I & II to see their association with Environmental Enteric Dysfunction.
Change in blood Low density lipoprotein related receptor 1 (LRP1) level | baseline and 3 months
  LRP1 is an endocytic receptor involved in trafficking at least 100 different molecules, including lipids and proteins/peptides involved in immune system function (e.g. antigen presentation) as well as viral proteins and toxins. The epigenetic data strongly suggest that LRP1 expression is reduced in stunted children compared to controls.
Change in blood metabolomic profile | baseline and 3 months
  Gut inflammation is reflected in an altered serum metabolite profile; characterization of the metabolome can identify pathways and metabolite bio-markers that may be useful as a diagnostic for inflammation
Change in small intestinal bacterial overgrowth (SIBO) status | baseline and 3 months
  Small intestine bacterial overgrowth (SIBO) is measured noninvasively by a hydrogen breath test, where oral glucose is administered and an increase of hydrogen in the breath SIBO of at least 12 parts per million is detected. Traditionally, SIBO has been considered a secondary condition that develops in the setting of altered intestinal anatomy, slowed intestinal motility, or aberrant gastrointestinal function.

CONTACTS AND LOCATIONS:
Locations (1):
- Mirpur, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pierce R, Jan NJ, Kumar P, Middleton J, Petri WA, Marie C. Persistent dysbiosis of duodenal microbiota in patients with controlled pediatric Crohn's disease after resolution of inflammation. Sci Rep. 2024 Jun 3;14(1):12668. doi: 10.1038/s41598-024-63299-y. PMID 38830904
- [Derived] Hossain MS, Begum SMKN, Rahman MM, Parvez M, Mazumder RN, Sarker SA, Hasan MM, Fahim SM, Gazi MA, Das S, Mahfuz M, Ahmed T. Environmental enteric dysfunction and small intestinal histomorphology of stunted children in Bangladesh. PLoS Negl Trop Dis. 2023 Jan 19;17(1):e0010472. doi: 10.1371/journal.pntd.0010472. eCollection 2023 Jan. PMID 36656867
- [Derived] Chen RY, Kung VL, Das S, Hossain MS, Hibberd MC, Guruge J, Mahfuz M, Begum SMKN, Rahman MM, Fahim SM, Gazi MA, Haque R, Sarker SA, Mazumder RN, Di Luccia B, Ahsan K, Kennedy E, Santiago-Borges J, Rodionov DA, Leyn SA, Osterman AL, Barratt MJ, Ahmed T, Gordon JI. Duodenal Microbiota in Stunted Undernourished Children with Enteropathy. N Engl J Med. 2020 Jul 23;383(4):321-333. doi: 10.1056/NEJMoa1916004. PMID 32706533
- [Derived] Mahfuz M, Alam MA, Das S, Fahim SM, Hossain MS, Petri WA Jr, Ashorn P, Ashorn U, Ahmed T. Daily Supplementation With Egg, Cow Milk, and Multiple Micronutrients Increases Linear Growth of Young Children with Short Stature. J Nutr. 2020 Feb 1;150(2):394-403. doi: 10.1093/jn/nxz253. PMID 31665385
- [Derived] Hossain MS, Das S, Gazi MA, Alam MA, Haque NMS, Mahfuz M, Ahmed T, Damman CJ. Association of faecal pH with childhood stunting: Results from a cross-sectional study. BMJ Paediatr Open. 2019 Sep 13;3(1):e000549. doi: 10.1136/bmjpo-2019-000549. eCollection 2019. PMID 31646200
- [Derived] Mahfuz M, Das S, Mazumder RN, Masudur Rahman M, Haque R, Bhuiyan MMR, Akhter H, Sarker MSA, Mondal D, Muaz SSA, Karim ASMB, Borowitz SM, Moskaluk CA, Barratt MJ, Petri WA, Gordon JI, Ahmed T. Bangladesh Environmental Enteric Dysfunction (BEED) study: protocol for a community-based intervention study to validate non-invasive biomarkers of environmental enteric dysfunction. BMJ Open. 2017 Aug 11;7(8):e017768. doi: 10.1136/bmjopen-2017-017768. PMID 28801442